CLINICAL TRIAL: NCT07327632
Title: A Multi-Center, Open-Label, Phase 1 Study of IBI3026 in Participants With Locally Advanced, Unresectable or Metastatic Solid Tumors
Brief Title: This is a Multi-Center Study of IBI3026 in Participants With Locally Advanced, Unresectable or Metastatic Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Innovent Biologics Technology Limited (Shanghai R&D Center) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI3026A101
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI3026 (Experimental)
  Interventions: Drug: IBI3026

INTERVENTIONS:
Drug: IBI3026 — Recombinant anti-programmed death receptor-1 (PD-1) antibody fused with interleukin-12 (IL-12) bispecific molecule injection

SUMMARY:
This is a multicenter, open-label, phase I dose-escalation and expansion study of IBI3026 in participants with unresectable, locally advanced, or metastatic solid tumors. The study will be conducted in two phases: Phase 1 dose escalation and Phase 2 dose expansion. Safety will be monitored by the Safety Review Committee (SRC).

ELIGIBILITY:
inclusion criteria:

1. Participants must have the ability to understand and sign a written informed consent form for participation in this study, including all assessments and procedures specified in the protocol;
2. Male or female participants aged ≥18 years;
3. At least one measurable lesion as defined by RECIST v1.1 within 28 days prior to the first dose of IBI3026;
4. ECOG performance status of 0-1;
5. Life expectancy of at least 12 weeks at the start of treatment;
6. The screening period confirms that bone marrow and organ functions are good.
7. Male or female participants who are either of non-reproductive potential or agree to use at least one highly effective method of contraception during the study period (starting from screening or 2 weeks prior to first dosing, whichever comes first, and continuing until 6 months after the last dose of study drug);
8. Not amenable to curative surgical resection or definitive chemoradiotherapy.

Exclusion criteria:

1. Prior treatment with IL-12 class cytokines or IL-12 inhibitors;
2. Participation in any interventional clinical study other than observational (non-interventional) studies, or currently in the follow-up period of an interventional study;
3. Adverse reactions from prior anti-tumor therapies that have not resolved to Grade 0 or 1, or baseline levels, according to NCI CTCAE v5.0, prior to the first dose of study drug (exceptions include alopecia, fatigue, hyperpigmentation, or other conditions deemed without safety risk by the investigator);
4. Prior immune checkpoint inhibitor therapy associated with severe adverse reactions sufficient to compromise participant safety;
5. Known hypersensitivity, allergic reaction, or intolerance to IBI3026 or its excipients (refer to Investigator's Brochure).
6. Received major surgery (e.g., craniotomy, thoracotomy, or laparotomy, or other surgeries as determined by the investigator) within 4 weeks prior to the first dose of study drug, excluding core biopsy; or anticipated to undergo major surgery during the study period; or presence of serious non-healing wounds, trauma, ulcers, etc.
7. Known symptomatic central nervous system (CNS) metastases. Participants with asymptomatic CNS metastases (i.e., no neurological syndrome and metastatic lesion diameter ≤1.5 cm) or those with stable disease post-treatment as judged by the investigator may be considered under the following conditions: absence of midbrain, pons, cerebellum, meninges, medulla oblongata, or spinal cord involvement; clinically stable for at least 4 weeks prior to the first dose of study drug (stable on ≤1.5 mg/day dexamethasone or equivalent corticosteroid and baseline anticonvulsant therapy), with no clinically confirmed new or enlarging CNS lesions.
8. Tumor invasion into surrounding critical structures (e.g., mediastinal vessels, superior vena cava, trachea, esophagus, etc.) or at risk of gastrointestinal/respiratory fistula formation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | up to 2 years
Serious Adverse Event | up to 2 years
Maximum Tolerated Dose | up to 2 years
DLT(Dose-limiting Toxicity) | up to 2 years

SECONDARY OUTCOMES:
PK concentration: IBI3026 serum concentration | up to 2 years
Incidence and number of patients with ADA | up to 2 years
Incidence and number of patients with NAb | up to 2 years
ORR (Objective Response Rate) | up to 2 years
DoR(Duration of Response) | up to 2 years
DCR(Disease Control Rate) | up to 2 years
TTR(Time to Response) | up to 2 years
PFS(Progression-free Survival) | up to 2 years
OS(Overall Survival) | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China